CLINICAL TRIAL: NCT05953129
Title: Novel Predictors of Post Spinal Hypotension in Cesarean Sections: Evaluating Jugular Vein Collapsibility Index and Shock Indices
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Oguz Özakın, Anesthesiology and Reanimation Specialist, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 126
Record Dates: First submitted 2023-07-12; First posted 2023-07-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cesarean Section Complications; Regional Anesthesia Morbidity; Hemodynamic Instability; Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Right Jugular Vein Collapsibility Index — Ultrasonography will be used to evaluate the diameter of the jugular vein (minimum and maximum values) and carotid diameter. The jugular vein collapsibility index will be measured by the anesthesiologist using non-invasive ultrasonography. Jugular vein collapsibility index will be calculated using the measured diameters.

SUMMARY:
Jugular vein collapsibility index and shock indices (Shock index, Modified Shock Index, Diastolic Shock Index) may be useful in estimating post spinal hypotension in cesarean section operations. Evaluation on the accuracy and effectiveness of these indices can contribute to the early diagnosis and management of hypotension. The main purpose of this study is to evaluate the effectiveness of shock indices in predicting the possibility of post spinal hypotension in cesarean section operations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-45 who had a planned cesarean section and approved to participate in the study and to apply spinal anesthesia

Exclusion Criteria:

* Patients with Preeclampsia, Eclampsia, HELLP syndrome

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women between the ages of 18-45 who were scheduled for cesarean section and who gave consent to participate in the study and to apply spinal anesthesia will be included in this study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Prediction of hypotension | 15 min
  To evaluate the ability of the jugular vein collapsibility index and shock indices (Shock index, Modified Shock Index, Diastolic Shock Index) to predict post spinal hypotension in cesarean section surgeries.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided